CLINICAL TRIAL: NCT03601208
Title: Comparison of Standard Venous Sampling for Measurement of Tacrolimus and Creatinine Versus Fingerprick Mitra® Volumetric Absorptive Microsampling in Adult Renal Transplant Recipients
Brief Title: Mitra v Fingerprick Tacrolimus Creatinine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18RE007
Record Dates: First submitted 2018-06-25; First posted 2018-07-26 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-06

CONDITIONS: Transplant;Failure,Kidney

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sample (Experimental): Venepuncture vs fingerprick test using Mitra volumetric absorptive microsampling (VAMs)
  Interventions: Diagnostic Test: Mitra

INTERVENTIONS:
Diagnostic Test: Mitra — When the patients have their bloods done through venepuncture, an additional 5-10mls will be taken (one EDTA bottle for tacrolimus and one serum bottle for creatinine; and two Mitra VAMs). Patients will also have a fingerprick test and 20 microlitres of blood taken using Mitra volumetric absorptive microsampling (VAMs)

SUMMARY:
Patients with kidney transplant have blood tests very often. This is normally done in hospital and using a needle inserted into the vein. Two tests are important for kidney transplant patients - creatinine to monitor the health of the kidney; and tacrolimus to measure the level of the medicine which prevents rejection. The investigators would like to compare a fingerprick microsampling method to the standard venous blood. The fingerprick test is the same done by patients with diabetes and we use a microsampling tip which looks like a cotton bud to draw up a small amount of blood. Each tip draws up exactly 10 microlitres which is two drops. The investigators want to compare the results of creatinine and tacrolimus done through the two methods. In the future, this would allow patients to do their creatinine and tacrolimus test at home. The tips dry completely and can be posted to a laboratory. We hope this will make life easier for transplant patients and also help them engage more with the care of their condition.

ELIGIBILITY:
Inclusion Criteria:

Kidney transplant recipients. Taking tacrolimus

Exclusion Criteria:

Unable to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of creatinine and tacrolimus values for Mitra VAM (test) versus venous sampling (standard). | 3 months
  Compare blood results for creatinine and tacrolimus using two different methods - Mitra volumetric absorptive microsamplers (VAM) versus venous blood (standard).

IPD SHARING:
Plan to Share IPD: No